CLINICAL TRIAL: NCT00472446
Title: Impact and Cost Efficiency of Bilateral, Superficial Cervical Block in Thyroid Surgery Under General Anesthesia
Brief Title: Superficial, Cervical Block in Thyroid Surgery, a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Thomas Steffen, attending surgeon, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EKSG 06/010/1B; 2006DR4184 (Other: SwissMedic)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Thyroidectomy
Keywords: Surgery; Thyroid gland; cervical block; Pain, Postoperative
MeSH Terms: conditions — Thyroid Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- cervical block before surgery (Experimental): bilateral superficial cervical block, placed before surgery (just before skin incision)
  Interventions: Drug: bilateral superficial cervical block
- placebo cervical block before surgery (Placebo Comparator): placebo bilateral superficial cervical block with saline, placed before surgery (just before skin incision)
  Interventions: Drug: placebo bilateral superficial cervical block
- cervical block after surgery (Experimental): bilateral superficial cervical block, placed after surgery (just after skin closure)
  Interventions: Drug: bilateral superficial cervical block
- placebo cervical block after surgery (Placebo Comparator): placebo bilateral superficial cervical block with saline, placed after surgery (just after skin closure)
  Interventions: Drug: placebo bilateral superficial cervical block

INTERVENTIONS:
Drug: bilateral superficial cervical block — 10 ml of 5% bupivacaine (Carbostesin®) was used for each side. Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
  Arms: cervical block after surgery; cervical block before surgery
Drug: placebo bilateral superficial cervical block — 10 ml of saline (the carrier of bupivacaine in the experimental treatment) was used for each side.
  Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
  Arms: placebo cervical block after surgery; placebo cervical block before surgery

SUMMARY:
The study investigates the impact on post-operative pain of the superficial cervical block with bupivacaine combined with subcutaneous infiltration of the incisional area in thyroid surgery under general anesthesia. In addition, cost savings using the cervical block are evaluated (due to reduced length of hospital stay).

The study is prospective, randomized, double blind, and placebo-controlled. The study is performed at the Department of Surgery, Cantonal Hospital of St. Gallen.

ELIGIBILITY:
Inclusion Criteria:

* Elective thyroid or combined thyroid/parathyroid surgery, restricted to the central cervical compartment
* Informed consent

Exclusion Criteria:

* Intolerance to used medication
* Recurrent disease
* Neck dissection, sternotomy
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clerici, MD, Principal Investigator — Department of Surgery, Cantonal Hospital St. Gallen
Locations (1):
- Department of Surgery, Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steffen T, Warschkow R, Brandle M, Tarantino I, Clerici T. Randomized controlled trial of bilateral superficial cervical plexus block versus placebo in thyroid surgery. Br J Surg. 2010 Jul;97(7):1000-6. doi: 10.1002/bjs.7077. PMID 20632263

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervivcal Block Before Surgery: bilateral superficial cervical block placed before surgery (just before skin incision)
  bilateral superficial cervical block: 10 ml of 5% bupivacaine (Carbostesin®) was used for each side.
  Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
- Cervivcal Block After Surgery: bilateral superficial cervical block placed after surgery (just after skin closure)
  bilateral superficial cervical block: 10 ml of 5% bupivacaine (Carbostesin®) was used for each side.
  Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
- Placebo Cervivcal Block Before Surgery: placebo bilateral superficial cervical block placed before surgery (just before skin incision)
  placebo bilateral superficial cervical block: 10 ml of saline (the carrier of bupivacaine in the experimental treatment) was used for each side.
  Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
- Placebo Cervivcal Block After Surgery: placebo bilateral superficial cervical block with saline placed after surgery (just after skin closure)
  placebo bilateral superficial cervical block: 10 ml of saline (the carrier of bupivacaine in the experimental treatment) was used for each side.
  Along the cranial dorsal edge of the sternocleidomastoid muscle, three deposits of approximately 2.5 ml were injected to anaesthetize the cervical plexus with its nervus transversus colli. To anaesthetize the region of the planned skin incision, the remaining 2·5 ml was injected subcutaneously on each side.
Period: Overall Study
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Started | 46 | 47 | 45 | 45
Completed | 41 | 41 | 38 | 39
Not Completed | 5 | 6 | 7 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Reintervention | 0 | 0 | 1 | 1
Not completed — Questionnaires not returned | 5 | 6 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery | Total
Number analyzed (Participants) | 41 | 41 | 38 | 39 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.0) | 46.5 (13.3) | 49.9 (13.5) | 47.3 (14.4) | 48.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 29 | 31 | 129
  Male | 8 | 5 | 9 | 8 | 30
Region of Enrollment [Number; unit: participants]
  Switzerland | 41 | 41 | 38 | 39 | 159
resection location [Number; unit: participants]
  unilateral | 18 | 22 | 24 | 26 | 90
  bilateral | 23 | 19 | 14 | 13 | 69
duration of surgery [Mean (Standard Deviation); unit: minutes] | 140.8 (48.1) | 130.5 (37.0) | 129.6 (48.1) | 141.9 (50.4) | 135.7 (45.7)
specimen weight [Mean (Standard Deviation); unit: gram] | 60.4 (55.1) | 42.2 (32.0) | 51.0 (43.6) | 39.8 (41.2) | 47.0 (43.4)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Measured by Visual Analogue Scale
Description: Patient administered Instrument to indicate pain on a level from 0 to 10. (0: no pain, 10: worst imaginable pain)
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
units on a scale | 2.15 (2.17) | 2.02 (2.06) | 2.84 (1.75) | 2.72 (1.89)
Statistical Analysis 1: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: no difference in outcome measure between superficial cervical block and placebo treatment (irrespective of timing of treatment); Test type: Superiority or Other; p = .028, t-test, 2 sided

2. Primary Outcome: Pooled Relative Treatment Effect of VAS
Description: Pain was obtained using the visual analog scale (VAS) three times daily for the 4 postoperative days (0 = no pain, 10 = worst imaginable pain)
  The pooled relative treatment effect is the probability of values being higher in one group than in another group (ranging from 0 to 1)
Time Frame: 4 days after surgery
Measure: Number (95% Confidence Interval); unit: pooled relative treatment effect
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
pooled relative treatment effect | 0.47 [0.43 to 0.51] | 0.45 [0.41 to 0.48] | 0.55 [0.51 to 0.59] | 0.54 [0.51 to 0.58]
Statistical Analysis 1: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.016, Non-parametric ANOVA-type statistic; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model
Statistical Analysis 2: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery; null hypothesis: no difference in outcome measure pre-operative versus post-operative application; Test type: Superiority or Other; p = 0.723, Non-parametric ANOVA-type statistic; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model

3. Secondary Outcome: Post-operative Pain Measured by Visual Analogue Scale
Description: Patient administered Instrument to indicate pain on a level from 0 to 10. (0: no pain, 10: worst imaginable pain)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
units on a scale | 1.95 (1.55) | 1.51 (1.48) | 2.20 (1.66) | 2.06 (1.39)

4. Secondary Outcome: Consumption of Post-operative Analgetics
Description: number of participants taking post-operative analgetics
Time Frame: 5 days after surgery
Measure: Number; unit: participants
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
participants
  paracetamol | 21 | 23 | 18 | 24
  metamizole | 6 | 7 | 3 | 7
Statistical Analysis 1: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: outcome measure (Proportion of patients taking analgetics) is equal between superficial cervical block and placebo treatment (irrespective of timing) Proportion taking Paracetamol:; Test type: Superiority or Other; p = 0.94, Fisher Exact; mid p value of the two-sided Fisher test
Statistical Analysis 2: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: outcome measure (Proportion of patients taking analgetics) is equal between superficial cervical block and placebo treatment (irrespective of timing) Proportion taking Metamizole:; Test type: Superiority or Other; p = 0.58, Fisher Exact; mid p value of two-sided Fisher test

5. Secondary Outcome: Mean Consumption of Post-operative Analgetics
Description: mean pooled dose of post-operative analgetics
Time Frame: 5 days after surgery
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
gram
  paracetamol | 3.33 (2.43) | 3.37 (2.43) | 4.06 (3.19) | 4.33 (3.56)
  metamizole | 1.25 (0.88) | .93 (0.61) | 2.46 (2.53) | 1.21 (0.64)
Statistical Analysis 1: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: no difference in pooled dose of analgetics, superficial block versus Placebo outcome: paracetamol; Test type: Superiority or Other; p = 0.328, Non-parametric ANOVA-type; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model
Statistical Analysis 2: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: no difference in pooled dose of analgetics, superficial block versus Placebo outcome: metamizole; Test type: Superiority or Other; p = 0.81, Non-parametric ANOVA-type; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model
Statistical Analysis 3: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery; null hypothesis: no difference in outcome measure pre-operative and post-operative application outcome measure: pooled paracetamol dose; Test type: Superiority or Other; p = 0.331, Non-parametric ANOVA-type statistic; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model
Statistical Analysis 4: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery; null hypothesis: no difference in outcome measure pre-operative and post-operative application outcome measure: pooled metamizole dose; Test type: Superiority or Other; p = 0.440, Non-parametric ANOVA-type statistic; Non-parametric ANOVA-type statistic for pooled main effects with Box approximation, full model

6. Secondary Outcome: Hospital Stay
Description: time from surgery to Hospital release in days
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Number analyzed (Participants) | 41 | 41 | 38 | 39
days | 1.8 (0.7) | 1.6 (0.7) | 2.0 (1.1) | 1.6 (0.6)
Statistical Analysis 1: Comparison: Cervivcal Block Before Surgery vs Cervivcal Block After Surgery vs Placebo Cervivcal Block Before Surgery vs Placebo Cervivcal Block After Surgery; null hypothesis: no difference in outcome measure for superficial cervical block versus placebo treatment; Test type: Superiority or Other; p = 0.925, non-parametric ANOVA-type statistic; non-parametric ANOVA-type statistic for pooled main effects, full model

ADVERSE EVENTS:
Time Frame: 6 weeks after surgery
Arm/Group | Cervivcal Block Before Surgery | Cervivcal Block After Surgery | Placebo Cervivcal Block Before Surgery | Placebo Cervivcal Block After Surgery
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/38 | 1/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/38 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervivcal Block Before Surgery (N=41) | Cervivcal Block After Surgery (N=41) | Placebo Cervivcal Block Before Surgery (N=38) | Placebo Cervivcal Block After Surgery (N=39)
hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes